CLINICAL TRIAL: NCT02093988
Title: Topical Tranexamic Acid in Major Paediatric Spine Deformity Surgery: A Randomized Controlled Trial
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H14-00595
Record Dates: First submitted 2014-03-18; First posted 2014-03-21 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Spinal Deformity, Paediatric Surgery, Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Topical and Intravenous TXA (Experimental)
  Interventions: Drug: Topical TXA; Drug: Intravenous TXA
- Intravenous TXA only (Active Comparator)
  Interventions: Drug: Intravenous TXA

INTERVENTIONS:
Drug: Topical TXA
  Other Names: TXA
  Arms: Topical and Intravenous TXA
Drug: Intravenous TXA
  Other Names: TXA

SUMMARY:
Our study will evaluate the use of topical and intravenous (IV) Tranexamic Acid (TXA) in spine surgery. The purpose of TXA is to prevent clotting during surgery to reduce blood loss. When used intravenously, it has been shown to safe, efficacious, and effective in reducing transfusion requirements and blood loss in spine surgeries. We want to evaluate the effect of using TXA topically and intravenously to see if it further reduces blood loss in children undergoing major surgery compared to IV TXA only

DETAILED DESCRIPTION:
Blood loss during major paediatric spine surgery is significant, and it is well established that patients undergoing such surgery have a substantial risk for requiring a blood transfusion in the perioperative period (1-4). Given the cost and associated risks with allogeneic blood product transfusion (5-7), a significant effort has been directed towards reducing transfusion requirements through various methods of blood conservation (8-12).

Tranexamic acid (TXA) is a synthetic antifibrinolytic that functions through competitive blockade of the lysine-binding sites of plasminogen, plasmin, and tissue plasminogen activator resulting in the inhibition of fibrinolysis and clot degradation (13). When used parentally, it has been shown to safe, efficacious, and effective in reducing transfusion requirements and blood loss during the perioperative period of various orthopaedic procedures, including major surgeries of the spine (14-23). A growing body of literature has supported the topical application of TXA in lower extremity joint reconstruction, among other procedures (24-29), in which a saline solution containing TXA is placed directly in the surgical incision prior to closure. Two randomized controlled trials have compared topical TXA and placebo for use in lumbar fusion and laminectomy cases. Both of these trials demonstrated a significant reduction in perioperative blood loss with the use of topical TXA as compared to placebo, and no reported no adverse events (36, 37).

While intravenous TXA has proven efficacy in reducing perioperative blood loss, despite its routine use during major paediatric spine surgery, blood loss and transfusion requirements remain significant (14-23). Thus, methods to further reduce perioperative blood loss in the children are of clinical significance. As highlighted above, topical TXA has clearly demonstrated excellent local anti-fibrinolytic action. Furthermore, when applied within a surgical incision, there is a negligible increase in serum TXA concentration (33-35).

We therefore propose a randomized trial to evaluate the effect of topical TXA on perioperative blood loss when used in addition to intravenous TXA for major paediatric spine surgery. In doing so, we seek to evaluate whether additional benefit may be conferred through direct application of TXA within the incision intravenous to that already provided by IV TXA. To date, such a question has not been evaluated in the surgical literature.

ELIGIBILITY:
Inclusion Criteria:

* All participants between ages of 8 and 21 years old
* All patients undergoing spinal deformity surgery for which operative time is anticipated to be greater than 3 hours - Operative time will be defined as time from incision to closure

Exclusion Criteria:

* Violation of the dura intraoperatively
* Requirement of therapeutic anticoagulation in the perioperative period
* Baseline coagulation disorder
* History of thromboembolic event, including, but not limited to:
* Myocardial infarction within past 6 months
* Deep vein thrombosis
* Pulmonary embolus
* Cerebrovascular accident or transient ischemic event
* Retinal artery occlusion
* Renal impairment - eGFR < 60 mL/min/1.73m2
* Pregnant
* Allergy to tranexamic acid
* Additional surgical procedures or interventions within the 7 days prior to the index spinal surgery, or within 72h following the index spinal surgery
* Planned staged procedures and procedures with less than 50 cc of blood loss not considered reason for study exclusion - Eg. change of negative pressure wound dressing, tracheostomy, central-line placement
* Inability of patient or legal guardian to provide study consent

Ages: 8 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 160 (Estimated)
Dates: Start 2015-08; Primary Completion 2017-02 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Volume of Blood Loss | Intra-operative

SECONDARY OUTCOMES:
Complications (reporting) | 6 week visit
  Any complications related to TXA administration will be recorded at the 6 week visit

CONTACTS AND LOCATIONS:
Overall Officials: Brett Kilb, Md, Study Chair — Resident; Firoz Miyanji, MD, Principal Investigator — Clinical Assistant Professor
Locations (1):
- BC Children's Hospital, Vancouver, British Columbia, Canada